CLINICAL TRIAL: NCT00532610
Title: A Randomized, Double-blind, Placebo-Controlled, Cross-Over Trial to Investigate the Effect of GSK189075 on Cardiac Repolarization as Compared to Placebo and a Single Dose of Moxifloxacin in Healthy Adult Subjects
Brief Title: A Study to Compare the Effect on Heart Rhythm of 3 Days of GSK189075, Placebo, or Moxifloxacin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KG2107489
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: Diabetes,; ECG,; Healthy Volunteers; GSK189075,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK189075

SUMMARY:
This study assesses for change in heart rhythm of healthy volunteers taking GSK189075 for 3 days at a normal dose and a higher than normal dose compared to placebo or to a single dose of moxifloxacin. Treatments are GSK189075 500mg daily for three days plus moxifloxacin placebo on Day 3; GSK189075 4000mg daily for three days plus moxifloxacin placebo on Day 3; placebo tablets daily for three days plus moxifloxacin placebo on Day 3; placebo tablets daily for three days plus Moxifloxacin 400mg on Day 3. Volunteers are blindfolded during dosing. Each volunteer participates in all four treatment periods and will have received each dose combination at study end. Volunteers will stay at the research unit from the day before the first dose of study drug until the day after the last dose of study drug of each period. Safety measures include vital signs, laboratory tests on blood and urine, physical exams and ECGs. Volunteers wear a Holter monitor (a device that records heart rate and rhythm continuously) on days 1 and 3. Study drug levels are assessed by multiple blood draws, most of which occur on day 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating females between 18 and 50 years of age (inclusive), at the time of signing the informed consent form.
* Body mass index (BMI) in the range of 19 to 32 (inclusive)
* Healthy as determined by a qualified physician on the basis of a satisfactory medical evaluation.
* Negative serum pregnancy test for all female subjects.
* Subject has given informed consent to participate in the study as indicated by providing a signed and dated written informed consent form prior to any study procedures.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Cardiac conduction and repolarization abnormalities described in the protocol.
* Any history of myocardial infarction, syncope, or cardiac arrhythmias or a history of uncontrolled hypertension or unstable heart disease.
* Subjects with a systolic blood pressure outside the range of 90 to 150mmHg or diastolic blood pressure outside the range of 50 to 100mmHg, or a greater than30mmHg change in systolic blood pressure or greater than 20mmHg change in diastolic blood pressure upon orthostatic vital signs.
* Subjects with a personal or family history of QTc prolongation or unexplained cardiac arrest.
* Liver function studies (ALT, AST, Total bilirubin, and alkaline phosphatase above 2 X the upper limit of the normal reference range at Screening and Day -2.
* Has a history of illicit drug use or alcohol abuse within the past year or a positive test for alcohol, cotinine, or drugs of abuse at Screening or prior to the start of dosing in Period 1.
* A history of regular alcohol consumption averaging >7 drinks/week for females or >14 drinks/week for males within 6 months of Screening.
* Use of tobacco or nicotine-containing products within 6 months prior to Screening and during the course of the study is prohibited.
* A positive test at Screening for Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV). If documented negative test results have been obtained within the last 2 months, it will not be necessary to repeat these tests.
* Any abnormalities of K+, Ca++ and Mg++
* TSH levels outside the normal range.
* Use of any prescription or non-prescription drugs, vitamins herbal and dietary supplements within fourteen days or 5 half-lives (whichever is longer) prior to the first dose of study drug. Drugs known to inhibit or induce CYP3A4 enzymes are restricted.
* Females of child-bearing potential who are unwilling or unable to use appropriate contraception as defined in the protocol.
* Pregnant or nursing females.
* Females who are using any oral contraception, implants of levonorgestrel, or injectable progesterone.
* Subjects whose participation in the study would result in donation of blood in excess of 500mL within a 56 day period.
* History of hypersensitivity to GSK189075, moxifloxacin, or drugs of these classes, or history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Continuous holter monitor & ECG each treatment period: | Days 1 & 3

SECONDARY OUTCOMES:
Drug plasma levels each treatment period: | Days 2 & 3
Safety ECG, labs, vital signs & adverse events: | each treatment period & follow-up
Day 3 change from baseline in QTcB, QTci, QT, and HR.
Blood drug levels of GSK189075 (pro-drug), GSK189074 (active entity), GSK279782 (active metabolite), GSK333081 (metabolite; may be analyzed as indicated by data from the dose escalation study) and moxifloxacin.
12-lead ECGs, vital signs, adverse events, and clinical laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States